CLINICAL TRIAL: NCT01821131
Title: A Dose Response, Randomized, Controlled, Double-blind, Cross-over Trial to Determine the LDL Cholesterol Lowering Effect of Ground Flaxseed in Adults With Above Optimal Plasma LDL Concentrations
Brief Title: Flax Muffins and Cholesterol Lowering
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B2013:012; RRC/2013/1281 (Other: Research Review Committee)
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Above Optimal Plasma LDL Concentrations
Keywords: flax; muffin; cholesterol; lignan; ALA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 30g ground flaxseed per day (Experimental): consume 1 muffin containing 30g ground flaxseed every day for 4 weeks
  Interventions: Other: muffin
- 20g ground flaxseed per day (Experimental): consume 1 muffin containing 20g ground flaxseed every day for 4 weeks
  Interventions: Other: muffin
- 0g ground flaxseed per day (Placebo Comparator): consume 1 muffin containing 0g ground flaxseed every day for 4 weeks
  Interventions: Other: muffin

INTERVENTIONS:
Other: muffin

SUMMARY:
This Clinical Trial is being conducted to study the LDL (bad) cholesterol lowering abilities of flax. The purpose of this study is to find the lowest dose of flax that can lower LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* male and non-pregnant/non-lactating female
* Body mass index 18.5-40.0 kg/m2
* Fasting plasma LDL cholesterol 2.6-5.0 mmol/L
* Regular dietary habits (ie. breakfast, lunch and dinner meals consumed daily)
* Willing to comply with protocol requirements
* Willing to provide informed consent

Exclusion Criteria:

* Medical history of cardiovascular disease, use of cholesterol-lowering or blood pressure-lowering medications
* Fasting plasma triglycerides ≥ 4.0 mmol/L
* Medical history of diabetes mellitus, fasting plasma glucose ≥ 7.0 mmol/L or use of insulin or oral medication to control blood sugar
* Medical history of gastrointestinal disease, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use within the past 6 weeks
* Medical history of inflammatory disease (ie. Systemic lupus erythematosis, rheumatoid arthritis, psoriasis)
* Medical history of liver disease or liver dysfunction (defined as plasma AST or ALT ≥ 1.5 times the upper limit of normal (ULN))
* Medical history of kidney disease or kidney dysfunction (defined as blood urea nitrogen and creatinine ≥ 1.8 times the ULN)
* Active treatment for any type of cancer within 1 year prior to study start
* Major surgery within the last 3 months
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
* Unstable body weight (defined as > 5% change in 3 months) or actively participating in a weight loss program
* Tobacco and/or nicotine replacement use, current or within the last 3 months
* Taking medication (prescription or non-prescription) or dietary supplements (pre/probiotics, vitamins, minerals, fats, herbals) known to affect blood lipids, with the exception of stable doses of thyroxine and oral contraceptive agents
* Any food allergy, aversion or unwillingness to eat wheat or flax
* Daily consumption of flax containing products in the past month
* Regular intake of > 2 alcoholic drinks per day. Standard drink (13.6 g alcohol)= Beer (5% alcohol) 360 mL (12 fl.oz); Spirits (40% alcohol) 45 mL (1.5 fl.oz); wine (12% alcohol) 150 mL (5 fl.oz)
* Participation in another clinical trial, current or in the past 4 weeks

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
lipid profile | 4 weeks
  plasma total cholesterol, HDL, LDL and triglycerides

SECONDARY OUTCOMES:
flax metabolites | 4 weeks
  plasma enterolignans and phospholipid fatty acid composition
blood pressure | 4 weeks
high sensitivity c-reactive protein (hsCRP) | 4 weeks
glucose | 4 weeks

OTHER OUTCOMES:
gastrointestinal side effects | 4 weeks
  participants will be asked to document any abnormal gastrointestinal side effects (ie. abdominal bloating/swelling, flatulence, constipation, diarrhea, stomach pain, nausea, belching, vomiting, chocking/difficulty swallowing)in their study diary.
liver function | 4 weeks
  plasma alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
kidney function | 4 weeks
  plasma creatinine and urea
Muffin acceptability questionnaire | 4 weeks
  Questionnaire evaluating how much the participants liked or disliked the muffins in terms of color, aroma, flavor, texture, overall acceptability and frequency of eating of the muffin after the study is complete. The questionnaire will be administered at the end of each phase after the participant has been consuming the muffin every day for 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada; Thomas Wolever, PhD, MD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Asper Clinical Research Institute, Winnipeg, Manitoba
  - Glycemic Index Laboratories Inc., Toronto, Ontario

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Genest J, McPherson R, Frohlich J, Anderson T, Campbell N, Carpentier A, Couture P, Dufour R, Fodor G, Francis GA, Grover S, Gupta M, Hegele RA, Lau DC, Leiter L, Lewis GF, Lonn E, Mancini GB, Ng D, Pearson GJ, Sniderman A, Stone JA, Ur E. 2009 Canadian Cardiovascular Society/Canadian guidelines for the diagnosis and treatment of dyslipidemia and prevention of cardiovascular disease in the adult - 2009 recommendations. Can J Cardiol. 2009 Oct;25(10):567-79. doi: 10.1016/s0828-282x(09)70715-9. PMID 19812802
- [Background] Charland SL, Cziraky MJ, Quimbo R, Karas RH, Insull W Jr, Davidson M, Stanek EJ. Achieving optimal lipid values in patients with dyslipidemia is associated with reduced risk of cardiovascular events. J Clin Lipidol. 2008 Oct;2(5):343-53. doi: 10.1016/j.jacl.2008.06.009. Epub 2008 Jun 26. PMID 21291759
- [Background] Lusis AJ. Atherosclerosis. Nature. 2000 Sep 14;407(6801):233-41. doi: 10.1038/35025203. PMID 11001066
- [Background] O'Rourke MF, Staessen JA, Vlachopoulos C, Duprez D, Plante GE. Clinical applications of arterial stiffness; definitions and reference values. Am J Hypertens. 2002 May;15(5):426-44. doi: 10.1016/s0895-7061(01)02319-6. PMID 12022246
- [Background] Xu Y, Wu Y, Li J, Ma W, Guo X, Luo Y, Hu D. The predictive value of brachial-ankle pulse wave velocity in coronary atherosclerosis and peripheral artery diseases in urban Chinese patients. Hypertens Res. 2008 Jun;31(6):1079-85. doi: 10.1291/hypres.31.1079. PMID 18716354
- [Background] Leng GC, Fowkes FG, Lee AJ, Dunbar J, Housley E, Ruckley CV. Use of ankle brachial pressure index to predict cardiovascular events and death: a cohort study. BMJ. 1996 Dec 7;313(7070):1440-4. doi: 10.1136/bmj.313.7070.1440. PMID 8973232
- [Background] Murabito JM, Evans JC, Larson MG, Nieto K, Levy D, Wilson PW; Framingham Study. The ankle-brachial index in the elderly and risk of stroke, coronary disease, and death: the Framingham Study. Arch Intern Med. 2003 Sep 8;163(16):1939-42. doi: 10.1001/archinte.163.16.1939. PMID 12963567
- [Background] Singh KK, Mridula D, Rehal J, Barnwal P. Flaxseed: a potential source of food, feed and fiber. Crit Rev Food Sci Nutr. 2011 Mar;51(3):210-22. doi: 10.1080/10408390903537241. PMID 21390942
- [Background] Bassett CM, Rodriguez-Leyva D, Pierce GN. Experimental and clinical research findings on the cardiovascular benefits of consuming flaxseed. Appl Physiol Nutr Metab. 2009 Oct;34(5):965-74. doi: 10.1139/H09-087. PMID 19935863
- [Background] Austria JA, Richard MN, Chahine MN, Edel AL, Malcolmson LJ, Dupasquier CM, Pierce GN. Bioavailability of alpha-linolenic acid in subjects after ingestion of three different forms of flaxseed. J Am Coll Nutr. 2008 Apr;27(2):214-21. doi: 10.1080/07315724.2008.10719693. PMID 18689552
- [Background] Zhang W, Wang X, Liu Y, Tian H, Flickinger B, Empie MW, Sun SZ. Dietary flaxseed lignan extract lowers plasma cholesterol and glucose concentrations in hypercholesterolaemic subjects. Br J Nutr. 2008 Jun;99(6):1301-9. doi: 10.1017/S0007114507871649. Epub 2007 Dec 6. PMID 18053310
- [Background] Othman RA, Moghadasian MH, Jones PJ. Cholesterol-lowering effects of oat beta-glucan. Nutr Rev. 2011 Jun;69(6):299-309. doi: 10.1111/j.1753-4887.2011.00401.x. PMID 21631511
- [Background] Bloedon LT, Balikai S, Chittams J, Cunnane SC, Berlin JA, Rader DJ, Szapary PO. Flaxseed and cardiovascular risk factors: results from a double blind, randomized, controlled clinical trial. J Am Coll Nutr. 2008 Feb;27(1):65-74. doi: 10.1080/07315724.2008.10719676. PMID 18460483
- [Background] Cunnane SC, Hamadeh MJ, Liede AC, Thompson LU, Wolever TM, Jenkins DJ. Nutritional attributes of traditional flaxseed in healthy young adults. Am J Clin Nutr. 1995 Jan;61(1):62-8. doi: 10.1093/ajcn/61.1.62. PMID 7825540
- [Background] Dodin S, Lemay A, Jacques H, Legare F, Forest JC, Masse B. The effects of flaxseed dietary supplement on lipid profile, bone mineral density, and symptoms in menopausal women: a randomized, double-blind, wheat germ placebo-controlled clinical trial. J Clin Endocrinol Metab. 2005 Mar;90(3):1390-7. doi: 10.1210/jc.2004-1148. Epub 2004 Dec 21. PMID 15613422
- [Background] Lucas EA, Wild RD, Hammond LJ, Khalil DA, Juma S, Daggy BP, Stoecker BJ, Arjmandi BH. Flaxseed improves lipid profile without altering biomarkers of bone metabolism in postmenopausal women. J Clin Endocrinol Metab. 2002 Apr;87(4):1527-32. doi: 10.1210/jcem.87.4.8374. PMID 11932276
- [Background] Patade A, Devareddy L, Lucas EA, Korlagunta K, Daggy BP, Arjmandi BH. Flaxseed reduces total and LDL cholesterol concentrations in Native American postmenopausal women. J Womens Health (Larchmt). 2008 Apr;17(3):355-66. doi: 10.1089/jwh.2007.0359. PMID 18328014
- [Background] Simbalista RL, Sauerbronn AV, Aldrighi JM, Areas JA. Consumption of a flaxseed-rich food is not more effective than a placebo in alleviating the climacteric symptoms of postmenopausal women. J Nutr. 2010 Feb;140(2):293-7. doi: 10.3945/jn.109.113886. Epub 2009 Dec 9. PMID 20007337
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- See also: Canadian health measures survey: Heart health and cholesterol levels of Canadians, 2007-2009 — http://www.statcan.gc.ca/pub/82-625-x/2010001/article/11136-eng.htm